CLINICAL TRIAL: NCT04528576
Title: Dragonfly-M Transcatheter Mitral Valve Repair System Early Feasibility Study
Brief Title: Dragonfly-M Early Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hangzhou Valgen Medtech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DragonFly-M-2020
Record Dates: First submitted 2020-08-23; First posted 2020-08-27 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2021-08

CONDITIONS: Mitral Regurgitation
Keywords: mitral regurgitation; TMVr
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: The clinical trial was designed as a single group assignment study. The participants with moderate to severe and severe mitral valve regurgitation will receive a transseptal mitral valve repair using Dragonfly mitral valve repair system.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DragonFly-M (Experimental): Experimental group is allocated to use novel mitral valve repair system manufactured by Hangzhou Valgen Meditech Co., Ltd
  Interventions: Device: Dragonfly mitral valve repair system

INTERVENTIONS:
Device: Dragonfly mitral valve repair system — With transesophageal echocardiographic guidance,implanting clip using Dragonfly mitral valve repair system

SUMMARY:
To establish the safety and effectiveness of the DragonFly transcatheter mitral valve repair system in symptomatic patients with moderate to severe and severe mitral regurgitation who have been determined to be at an high risk of mortality with mitral valve surgery by the cardiac surgeon with concurrence by the local Heart Team

DETAILED DESCRIPTION:
The subjects with moderate-to-severe (3+) and severe (4+) mitral valve regurgitation (MR) at high or prohibitive surgical risk will be evaluated by the study sites, and study eligibility confirmed by the echocardiographic core laboratory and eligibility committee. Those qualifying will then be treated with Dragonfly transcatheter mitral valve repair system after signing the informed consent. The follow-up will be conducted at discharge, 30 days, 6 months and 12 months after the operation. The primary endpoints are the incidence of major adverse events (MAE) at 30 days, and acute procedural success. Acute procedural success is defined as placement of one or more Dragonfly devices on the mitral valve with reduction of MR to 2+ or less. The secondary endpoints include all-cause mortality, cardiovascular mortality, incidence of serious adverse event, cardiovascular rehospitalization, NYHA functional class, mitral valve hemodynamics, acute technical success rate and device success rate at 6 months. Acute technical success is defined as no procedural mortality, successful in access, delivery, and retrieval of the device delivery system, and no emergency surgery or reintervention related to the device or access procedure in the catheterization laboratory. Device success is defined as no procedural mortality, proper delivery and deployment of the device, no unplanned surgical or interventional procedures related to the device, no specific device-related technical failure and or complications, function improvement of MR without significant stenosis (MR ≤ 2+) and without associated hemolysis or thrombogenesis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 yrs
2. Moderate-to-severe (3+) or severe (4+) mitral valve regurgitation on transthoracic or transesophageal echocardiography, and confirmed by echocardiographic core laboratory
3. The patient is on optimal guideline directed medical therapy for heart failure and remains symptomatic.
4. High or prohibitive surgical risk as defined by either Society for Thoracic Surgery Risk Calculator score for valve replacement ≥ 8 points; or STS score for valve repair ≥ 6 points , prohibitive risk as determined by the clinical judgement of the site heart team, including a cardiac surgeon experienced in mitral valve surgery and a cardiologist experience in mitral valve disease, due to the presence of one or more documented surgical risk factors.
5. Anatomically suitable for mitral valve repair and can be treated by Dragonfly confirmed by both site investigators, echocardiographic core laboratory, and the eligibility committee.
6. Transseptal catheterization and femoral vein access is determined to be feasible
7. Life expectancy ≥ 12 months
8. The subject or the subject's legal representative has been informed of the nature of the trial, willing to accept the experimental tests and follow-ups, and has provided written informed consent

Exclusion Criteria:

1. History of heart transplantation, prior mitral valve replacement surgery. or transcatheter mitral valve procedure;
2. Leaflet anatomy which may preclude Dragonfly-MTM implantation and position, as judged by the site investigators and confirmed by the echocardiographic core laboratory and eligibility committee
3. Evidence of calcification or significant cleft in the grasping area
4. LVEF < 20%
5. LVESD≥ 60mm;
6. Mobile leaflet length<10mm
7. Mitral valve effective orifice area (EOA) < 3.5cm2 or in the opinion of site investigators and confirmed by the echocardiographic core laboratory and eligibility committee that mitral stenosis would result from implantation of the Dragonfly-MTM device.
8. Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
9. Severe non-mitral valve disease requiring treatment .
10. Severe pulmonary artery hypertension (sPAP>70mmHg)
11. Severe right ventricular dysfunction;
12. Active endocarditis or previous mitral valve endocarditis; Active rheumatic heart disease or leaflets degenerated from rheumatic disease
13. Severe untreated coronary artery stenosis requiring revascularization; or with other cardiovascular disease requiring surgical treatment；
14. Extreme frailty
15. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis and any other structural heart disease causing heart failure other than dilated cardiomyopathy;
16. Renal failure requiring dialysis;
17. Blood cachexia including granulocytopenia (WBC < 3×109/L), acute anemia (HB < 90g/L), thrombocytopenia (PLT < 50×109/L), severe coagulopathy, and contradictions of anticoagulant and antiplatelet agents;
18. Evidence of an acute myocardial infarction in the prior 4 weeks;
19. Evidence of a shock in the prior 90 days;
20. Any percutaneous cardiac intervention or carotid surgery or any cardiac surgery within the 30 days prior to randomization;
21. Evidence of acute peptic ulcer upper or gastrointestinal hemorrhage in the prior 90 days;
22. Severe symptomatic carotid artery stenosis over 70% confirmed by echocardiography;
23. The subjects suffer from diseases which may lead difficulty in evaluating treatment (e.g., cancer, infection, severe metabolic disease, psychosis, etc.); or special cases that were evaluated by the heart team of local experimental center as not suitable for the surgical application of this clinical trial;
24. Life expectancy ≤ 12 months;
25. Subject participating in an investigational drug or another device study within the past 1 month;
26. In the judgment of the investigator, subjects may not complete the trial according to poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute procedural success | 1 month
  The acute procedural success is defined as successful Dragonfly implantation, and residual MR of 2+ or less at discharge. An echocardiogram at 30 days can be accepted if the discharge image was not available or hard to interpret. A death before discharge or a re-operation of mitral valve prior to 30 days is defined as acute procedure failure
Incidence of major adverse event (MAE) at 30 days | 1 month
  Major adverse event is defined as one of the following components: death, myocardial infarction (MI), stroke, renal failure requiring dialysis, and cardiac surgery for Dragonfly device failure.

SECONDARY OUTCOMES:
All-cause mortality | 6 months
  Death from any cause
Cardiovascular mortality | 6 months
  Death from cardiac causes
Incidence of serious adverse event (SAE） | 6 months
  If the adverse event meets any of the criteria below, it is regarded as a serious adverse event (SAE): 1) results in death; 2) is life threatening, results in illness or injury; 3) requires inpatient hospitalization or prolongation of existing hospitalization; 4) results in a persistent or significant disability/incapacity; 5) results in a congenital anomaly/birth defect, fetal death, fetal distress; 6) results in medical or surgical intervention to prevent permanent impairment to body structure or a body function; 7) an important medical event that may not result in death, be life-threatening, or require hospitalization but may be considered serious when, based upon appropriate medical judgment, may jeopardize the patient or subject and/or may require intervention to prevent one of the outcomes listed in this definition.
NYHA | 6 months
  NYHA functional class
Technical success | Immediately after procedure
  must meet all of the following items: 1) no procedural mortality; and 2) successful in access, delivery, and retrieval of the device delivery system; and 3) no emergency surgery or reintervention related to the device or access procedure.
Device success | 6 months
  must meet all of the following items:1) No procedural mortality; 2) Proper delivery and deployment of the device; 3) No unplanned surgical or interventional procedures related to the device; 4) No specific device-related technical failure or complication. 5) Improvement of MR without significant stenosis (MR ≤ 2+) without associated hemolysis or thrombogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: jianan Wang, PhD, Principal Investigator — Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu X, Chen M, Han Y, Pu Z, Lin X, Feng Y, Xu K, Lam YY, Lim DS, Wang J. First-in-Human Study of the Novel Transcatheter Mitral Valve Repair System for Mitral Regurgitation. JACC Asia. 2022 Jun 21;2(3):390-394. doi: 10.1016/j.jacasi.2022.03.010. eCollection 2022 Jun. PMID 36338402

DOCUMENTS (1):
  • Study Protocol (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/76/NCT04528576/Prot_000.pdf